CLINICAL TRIAL: NCT02446028
Title: A Randomized, Open-label Parallel Group Phase 2b Trial Evaluating Safety and Efficacy of BIOD 531 Compared to Humalog® Mix 75/25 in Subjects With Type 2 Diabetes
Brief Title: A Study Evaluating Safety and Efficacy of BIOD 531 Compared to Humalog® Mix 75/25 in Subjects With Type 2 Diabetes
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: IND Withdrawn
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-250
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIOD-531 (Experimental): BIOD-531 injected twice daily
  Interventions: Drug: BIOD-531
- Humalog® Mix 75/25 (Active Comparator): Humalog® Mix 75/25 injected twice daily
  Interventions: Drug: Humalog® Mix 75/25

INTERVENTIONS:
Drug: BIOD-531
  Arms: BIOD-531
Drug: Humalog® Mix 75/25
  Arms: Humalog® Mix 75/25

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BIOD-531 compared to Humalog®Mix 75/25 in patients with type 2 diabetes.

DETAILED DESCRIPTION:
BIOD-531 is a formulation of recombinant human insulin with a biphasic absorption profile characterized by rapid absorption (to prevent meal-time rises in blood glucose) and a secondary longer (basal) phase. The purpose of this trial is to evaluate glucose control and safety of BIOD-531 compared to a pre-mixed insulin which is commonly used to provide both meal-time and long acting insulin.

ELIGIBILITY:
Inclusion Criteria:

* Established clinical diagnosis of type 2 diabetes, consistent with ADA classification criteria for 6 months or longer.
* Body Mass Index 27 - 45 kg/square meter, inclusive.
* Screening HbA1c between 7.5 and 11.0%, inclusive.
* Up to two injections per day of U-100 basal (NPH, glargine, or detemir), pre-mixed, or self-mixed basal/prandial insulins or insulin analogs at stable total daily doses between 40 -200 units/day, inclusive, for ≥ 3 months prior to screening.

Exclusion Criteria:

* Regular use of Humulin®R U-500 or sulfonylurea, exenatide (short-acting), repaglinide, or nateglinide within 1 month prior to screening.
* History of bariatric surgery.
* Subject has had one or more severe hypoglycemic episodes associated with seizure, coma, or unconsciousness within the past 6 months.
* History of known hypersensitivity to any of the components in the study medication.
* New York Heart Association (NYHA) Class III or IV functional capacity, unstable angina pectoris, myocardial infarction, severe peripheral vascular disease, ischemic strokes or transient ischemic attacks within 6 months of screening.
* Systolic blood pressure ≥ 180 mmHg or sitting diastolic blood pressure ≥ 100 mmHg confirmed on repeat during screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 18 weeks

SECONDARY OUTCOMES:
Postprandial glucose excursions | 18 weeks
Change in weight | 18 weeks
Hypoglycemic event rates | 18 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Meridien Research, Bradenton, Florida
  - Endocrine Research Solutions, Roswell, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Springfield Diabetes and Endocrine Center, Springfield, Illinois
  - Diabetes and Endocrinology Consultants, Morehead City, North Carolina
  - Clinical Trials of Texas, San Antonio, Texas
  - Ranier Clinical Research Center, Renton, Washington